CLINICAL TRIAL: NCT00208546
Title: Cetuximab Added to Capecitabine, Oxaliplatin and Bevacizumab in Patients With Previously Untreated Advanced Colorectal Carcinoma, a Randomised Phase III Study
Brief Title: Cetuximab, Capecitabine, Oxaliplatin and Bevacizumab in Advanced Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dutch Colorectal Cancer Group (Other)
Collaborators: Koningin Wilhelmina Fonds (Other); Sanofi (Industry); Roche Pharma AG (Industry); Immunicon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIRO2
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer
Keywords: capecitabine; oxaliplatin; bevacizumab; cetuximab; advanced colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1Capecitabine + bevacizumab + oxaliplatin + cetuximab (Experimental)
  Interventions: Drug: 1Capecitabine + oxaliplatin + bevacizumab + cetuximab
- 21Capecitabine + bevacizumab + oxaliplatin (Active Comparator)
  Interventions: Drug: 21Capecitabine + bevacizumab + oxaliplatin

INTERVENTIONS:
Drug: 21Capecitabine + bevacizumab + oxaliplatin — 3-weekly cycles: Ca 1000 mg/m2 orally day 1-14, O 130 mg/m2 i.v. day 1 (6 cycles), B 7,5 mg/kg i.v. day 1.
  Arms: 21Capecitabine + bevacizumab + oxaliplatin
Drug: 1Capecitabine + oxaliplatin + bevacizumab + cetuximab — 3-weekly cycles: Ca 1000 mg/m2 orally day 1-14, O 130 mg/m2 i.v. day 1 (6 cycles), B 7,5 mg/kg i.v. day 1, Ce 250 mg/m2 i.v. day 1, 8, 15 (day 1 cycle 1: 400 mg/m2).
  Arms: 1Capecitabine + bevacizumab + oxaliplatin + cetuximab

SUMMARY:
This is a study to assess the efficacy and safety of the addition of cetuximab to the combined regimen of capecitabine, oxaliplatin and bevacizumab in patients with previously untreated advanced colorectal carcinoma. It is an open, comparative study, comparing the effects of capecitabine, oxaliplatin and bevacizumab to those of the same regimen plus cetuximab.

Seven hundred fifty patients will be included. Treatment will continue until disease progression or serious toxicity and follow up will continue until death. It is anticipated that the addition of cetuximab will lead to an increase in progression free survival.

DETAILED DESCRIPTION:
Primary objective: To assess the efficacy, defined as progression-free survival (PFS), of adding cetuximab to capecitabine/oxaliplatin/bevacizumab for advanced CRC.

Secondary objectives: To assess tumour response (CR, PR or SD), response duration, overall survival, toxicity profile, quality of life, translational research.

Methodology: Open, randomised multicenter phase III study. The number of patients is 750.

Test products: All cycles will be administered q 3 weeks. Oxaliplatin will be discontinued after 6 cycles in both study arms. The dose of capecitabine will be increased to 1250 mg/m2 b.i.d. as of cycle 7.

Arm A: capecitabine 1000 mg/m2 orally b.i.d. on day 1-14 (1250 mg/m2 after 6 cycles), oxaliplatin 130 mg/m2 i.v. infusion on day 1 during 6 cycles, bevacizumab 7.5 mg/kg i.v. infusion on day 1.

Arm B: capecitabine 1000 mg/m2 orally b.i.d. on day 1-14 (1250 mg/m2 after 6 cycles), oxaliplatin 130 mg/m2 i.v. infusion on day 1 during 6 cycles, bevacizumab 7.5 mg/kg i.v. infusion on day 1. Cetuximab 400 mg/m2 i.v. day 1 of cycle 1, thereafter weekly 250 mg/m2 i.v.

Duration of treatment and follow-up: Treatment is continued until disease progression, or unacceptable toxicity. Patients will be evaluated every 9 weeks for response while on treatment, or at any other time point when progression is suspected. After cessation of therapy for reasons other than disease progression, patients will be followed every 3 months until progression or death. Death and/or progression should be reported whenever it occurs.

In case chemotherapy (i.e. capecitabine and/or oxaliplatin) is discontinued for reasons of toxicity, treatment with bevacizumab (arm A) or bevacizumab + cetuximab (Arm B) should be continued until progression or unacceptable toxicity. Also, if chemotherapy plus bevacizumab is discontinued in Arm B for reasons of toxicity, treatment with cetuximab should be continued until progression or unacceptable toxicity.

Criteria for evaluation:

Efficacy: All eligible patients will be included in the analysis (intent-to-treat). All patients receiving > 9 weeks of treatment (i.e. 3 cycles) will be considered evaluable for response, unless documented progression occurred earlier.

Safety profile: Safety will be analysed in each treatment group. Patients having received ≥ 1 treatment doses are evaluable for toxicity. Evaluation will be performed on the safety population (having received treatment, assignment to treatment groups as treated). Clinical and laboratory toxicity/symptomatology will be graded according to NCI common toxicity criteria, version 3.0. The adverse events which are not reported in NCI common toxicity criteria will be graded as: mild, moderate, severe, life threatening.

Statistical methodology: The main endpoint of the study is the progression free survival interval (PFS). PFS curves will be constructed by means of the Kaplan Meier method. Comparisons of PFS curves will performed by mean of the log rank test. Similar methods will be used to analyse the duration of survival. All analyses will be done according to the intention-to-treat principle.

The expected median PFS in Arm A (standard arm) is 11 months. The minimum increase in PFS in Arm B (experimental arm) will be 3 months (21% hazard ratio reduction). 540 events are required for 80% power. 740 patients are needed to show this difference (>=0.05, 2-tailed test). To allow for ineligibility in some patients, a total of 750 patients will be included.

Stratification parameters:

Patients will be stratified for the following parameters:

* Prior adjuvant therapy (yes versus no);
* Number of organs affected (1 versus > 1, in case the primary tumour is in situ this will count as one organ);
* Serum LDH (normal versus above normal);
* Per participating institution.

Side studies: Side studies on prognostic factors in tumour samples from included patients will be performed, as well as on circulating tumour cells and endothelial cells and serum proteomics.

ELIGIBILITY:
Inclusion Criteria:

Histology and Staging Disease

* Histologically proven advanced colorectal cancer (CRC); not amenable to curative surgery
* Of Note: In case of a single metastasis, histological or cytological proof of colorectal carcinoma should be obtained prior to randomisation.
* Unidimensionally measurable disease (>= 1 cm on spiral CT scan or >= 2 cm on chest X-ray; liver ultrasound not allowed). Index lesions should not be in a previously irradiated area. Serum carcinoembryonic antigen (CEA) may not be used as a parameter for disease evaluation.
* In case of previous radiotherapy, at least one measurable lesion should be located outside the irradiated field.

General Conditions

* Signed written informed consent
* Age 18 years and above
* World Health Organization (WHO) performance status 0-1
* Adequate bone marrow function (white blood cell count [WBC] > 3.0 x 10^9/L, platelets > 100 x 10^9/L, hemoglobin [Hb] > 6 mmol/L)
* Adequate hepatic function: total bilirubin < 2 x upper normal limit, aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) < 3 x upper normal limits (in case of liver metastases < 5 x upper normal limits)
* Adequate renal function: serum creatinine < 1.5 x upper normal limit
* Urinary protein excretion < 0.5 gram/24h
* Expected adequacy of follow-up

Exclusion Criteria:

* Prior chemotherapy for advanced disease; prior adjuvant chemotherapy is allowed provided that the last administration was given > 6 months prior to randomisation, and that patients have recovered from all toxic events related to adjuvant chemotherapy, and that safety evaluations during adjuvant chemotherapy do not present any risk for serious adverse events during the administration of protocol treatment.
* Previous radiotherapy for rectal cancer or for symptomatic treatment of distant metastases is allowed, provided that at least one measurable lesion is located outside the irradiated field, irradiation has been completed for at least 4 weeks, and patients have recovered from all side effects.
* Previous epidermal growth factor receptor (EGFR) targeting therapy
* Sensory neuropathy > grade 1
* Bleeding diathesis or coagulation disorders or the need for full-dose anticoagulation
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the start of drug administration
* Anticipated major surgical procedure during the course of the study
* Serious non-healing wound or ulcer
* Any condition preventing the intake or absorption of oral drugs
* Significant cardiovascular disease (unstable angina pectoris, recent myocardial infarction < 12 months, uncontrolled hypertension, previous cerebrovascular disease)
* Pregnancy or lactation
* Patients (males/females) with reproductive potential not implementing adequate contraceptive measures
* Central nervous system metastases (in asymptomatic patients no screening is required)
* Serious active infections
* Other serious concomitant diseases preventing the safe administration of study drugs or likely to interfere with the study assessments
* Other malignancies in the past 5 years with the exception of adequately treated carcinoma in situ of the cervix or squamous or basal cell carcinoma of the skin
* Concomitant treatments: concomitant (or within 4 weeks before randomisation) administration of any other experimental drug under investigation; concurrent treatment with any other anti-cancer therapy; full-dose anticoagulation
* Continuous use of immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2005-06; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
progression free survival | study duration
toxicity | study duration

SECONDARY OUTCOMES:
tumour response (complete response [CR], partial response [PR] or stable disease [SD]) | study duration
response duration | study duration
overall survival | study duration
quality of life | study duration
translational research | study duration

CONTACTS AND LOCATIONS:
Overall Officials: C JA Punt, MD PhD, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Center Nijmegen, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] Tol J, Koopman M, Rodenburg CJ, Cats A, Creemers GJ, Schrama JG, Erdkamp FL, Vos AH, Mol L, Antonini NF, Punt CJ. A randomised phase III study on capecitabine, oxaliplatin and bevacizumab with or without cetuximab in first-line advanced colorectal cancer, the CAIRO2 study of the Dutch Colorectal Cancer Group (DCCG). An interim analysis of toxicity. Ann Oncol. 2008 Apr;19(4):734-8. doi: 10.1093/annonc/mdm607. Epub 2008 Feb 13. PMID 18272912
- [Result] Tol J, Koopman M, Cats A, Rodenburg CJ, Creemers GJ, Schrama JG, Erdkamp FL, Vos AH, van Groeningen CJ, Sinnige HA, Richel DJ, Voest EE, Dijkstra JR, Vink-Borger ME, Antonini NF, Mol L, van Krieken JH, Dalesio O, Punt CJ. Chemotherapy, bevacizumab, and cetuximab in metastatic colorectal cancer. N Engl J Med. 2009 Feb 5;360(6):563-72. doi: 10.1056/NEJMoa0808268. PMID 19196673
- [Derived] Baas J, Krens L, Bohringer S, Mol L, Punt C, Guchelaar HJ, Gelderblom H. Genome wide association study to identify predictors for severe skin toxicity in colorectal cancer patients treated with cetuximab. PLoS One. 2018 Dec 17;13(12):e0208080. doi: 10.1371/journal.pone.0208080. eCollection 2018. PMID 30557370
- [Derived] van Kessel CS, Samim M, Koopman M, van den Bosch MA, Borel Rinkes IH, Punt CJ, van Hillegersberg R. Radiological heterogeneity in response to chemotherapy is associated with poor survival in patients with colorectal liver metastases. Eur J Cancer. 2013 Jul;49(11):2486-93. doi: 10.1016/j.ejca.2013.03.027. Epub 2013 May 18. PMID 23692811
- [Derived] Simkens LH, Koopman M, Mol L, Veldhuis GJ, Ten Bokkel Huinink D, Muller EW, Derleyn VA, Teerenstra S, Punt CJ. Influence of body mass index on outcome in advanced colorectal cancer patients receiving chemotherapy with or without targeted therapy. Eur J Cancer. 2011 Nov;47(17):2560-7. doi: 10.1016/j.ejca.2011.06.038. Epub 2011 Jul 29. PMID 21803570
- See also: Related Info — http://www.dccg.nl